CLINICAL TRIAL: NCT00414882
Title: A Cluster-Randomized Trial of DOTS Versus DOTS Plus Active Case Finding to Reduce Tuberculosis Incidence in Rio de Janeiro, Brazil
Brief Title: A Cluster-Randomized Trial of DOTS vs DOTS Plus Active Case Finding
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 06-0017
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2011-04

CONDITIONS: Mycobacterium Tuberculosis
Keywords: TB, tuberculosis, Mycobacterium tuberculosis, Brazil
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of the study is to see if one plan for identifying and treating tuberculosis (TB) works better than another in reducing new cases of TB. The first plan is the DOTS program, which provides free TB treatment to people seeking it. The second plan provides free TB treatment to people seeking it and involves program staff going door-to-door in communities to identify new cases of TB, DOTS plus active case-finding program (ACF). Researchers believe that by detecting TB cases earlier and supervising treatment it will help to prevent spreading and decrease TB in these areas. The study population will be 200,000 people in 6 communities of Santa Cruz and 14 communities of Northeast Rio de Janeiro, Brazil, receiving DOTS or DOTS plus ACF. Individuals in the DOTS plus ACF part of the study will be interviewed 2-4 times during a 9 month period. Patients with symptoms will provide a sputum specimen. Patients identified as having TB will begin treatment and be observed for 6.

DETAILED DESCRIPTION:
Tuberculosis (TB) continues to be a major cause of morbidity and mortality worldwide, particularly in developing countries. The World Health Organization (WHO) has estimated that one-third of the world's population is infected with Mycobacterium tuberculosis. Tuberculosis remains a major public health problem in Brazil, being the 15th highest TB burden in the world. The goal of this project is to determine whether TB active case finding (ACF) in conjunction with directly observed therapy (DOTS) results in lower incidence of TB compared with routine DOTS alone. This community-randomized trial will be conducted in 20 Rio de Janeiro communities within 2 APs with high rates of TB where community health workers and health units are undergoing intensive training to implement DOTS programs. This will be a collaborative effort between the Municipal Health Secretariat of Rio de Janeiro and the Johns Hopkins University Center for Tuberculosis Research. A cluster-randomized trial will be conducted to compare the impact of 2 case detection and treatment strategies on the community incidence of TB. The 20 communities within 2 planning areas (APs) will be randomly assigned to routine DOTS based on passive case detection or DOTS+ACF, where TB cases are actively detected by community outreach. In all communities, cases of TB will be identified through the existing TB clinics using identical procedures for subjects reporting to the TB clinics on their own accord. These subjects will be identified through traditional methods of passive case finding (PCF). In DOTS+ACF communities, all households will be surveyed by community health workers to identify individuals with cough for greater than or equal to 3 weeks, and all symptomatic subjects will provide a spot sputum specimen for acid-fast bacilli smear at the time of their household survey. Results will be returned to the subject at their home and appropriate follow-up measures will be provided to confirm TB diagnoses and provide treatment. The primary objective of the study is to compare TB incidence in communities randomized to DOTS+ACF and DOTS alone over the 18-month period following ACF campaign. The study hypothesizes that the average TB incidence in these 18 months will be 42% less in the DOTS+ACF arm compared with the DOTS-arm. The study has two secondary objectives. The first secondary objective will be to compare case notification rates of TB in the 2 arms of the study during the ACF campaign. Researchers hypothesize that TB notification rates will be at least 40% greater in the DOTS+ACF communities during the ACF period of the study. The second secondary objective will be to compare treatment completion rates between the 2 arms of the study. Researchers hypothesize that subjects detected through ACF will have equal treatment completion rates (+/- 5%) as subjects in the DOTS-arm. Tuberculosis diagnosis is the primary outcome measure. Treatment completion is the secondary outcome measure. The study population will be residents of the 20 communities selected, approximately 200,000 people with no restriction on age. Diagnosing subjects earlier will ensure that they are treated earlier and have less time to spread the disease to their contacts.

ELIGIBILITY:
Inclusion Criteria:

All residents of the study communities will be eligible to be surveyed at their homes, regardless of gender, age, or ethnicity. In the DOTS+ACF communities, all households will be surveyed and symptomatic subjects will provide sputum specimens. The subjects will be males and females with no restriction on age, with and without active TB, and living in communities with a high prevalence of TB.

There will be no exclusion of women or minorities in this study. Pregnant women will be included if they have TB or live in a household with a TB case.

Children will be included if they have TB per routine practice and will be surveyed in the DOTS+ACF arm for symptoms with their parent's verbal permission and presence.

Exclusion Criteria:

All residents of the 20 selected communities will be eligible to participate in the study. Consent will not be requested for DOTS, because this is now the standard of care for the area. Verbal consent will be requested for use of household data to analyze the effectiveness of active case finding. However, even households that refuse to participate in the survey (which is extremely unlikely because this is part of the routine survey in which all households currently participate) will be included when calculating TB incidence for the community.

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200000
Dates: Start 2007-07-10; Primary Completion 2009-06-28 (Actual); Study Completion 2012-06

CONTACTS AND LOCATIONS:
Locations (1):
- Municipal Health Department, Rio de Janeiro, Brazil